CLINICAL TRIAL: NCT03383926
Title: Prospective Study About the Efficacy of the Longo's Intervention for the Treatment of Hemorrhoids and Rectal Mucosal Prolapse.
Brief Title: Longo's Intervention in the Treatment of Hemorrhoids and Rectal Mucosal Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Mataró (Other)
Responsible Party: Principal Investigator, Luis Antonio Hidalgo Grau, MD, PhD, Hospital de Mataró
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LONGO
Record Dates: First submitted 2017-09-12; First posted 2017-12-27 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Hemorrhoids; Rectal Mucosa Prolapse
Keywords: Longo; Hemorrhoids; Rectal; Prolapse; Anal
MeSH Terms: conditions — Hemorrhoids; Rectal Prolapse; Prolapse | interventions — Sutures

STUDY DESIGN:
Intervention Model Description: In the surgery, Longo's intervention would be done by two ways differing in the distance of the suture from the tobacco pouch to the anal margin (4.5 cm in the first group and 6 cm in the second group).
Who Masked: Participant, Outcomes Assessor
Masking Description: Neither the evaluator of the research and the participant do not know the lenght of the Longo's intervention that is performed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Suture confection of theTobacco-pouch of 4.5cm from the anal margin.
  Interventions: Procedure: 4.5cm suture
- Group 2 (Experimental): Suture confection of theTobacco-pouch of 6cm from the anal margin.
  Interventions: Procedure: 6cm suture

INTERVENTIONS:
Procedure: 4.5cm suture — Suture confection of the Tobacco-pouch of 4.5cm from the anal margin.
  Arms: Group 1
Procedure: 6cm suture — Suture confection of the Tobacco-pouch of 6cm from the anal margin.
  Arms: Group 2

SUMMARY:
The aim of this study is to define the significance of the distance of the staple line to the dentate line of the anal canal in the efficacy of the Longo's intervention.

DETAILED DESCRIPTION:
Is going to be carried out with patients from 18 to 70 years old with hemorrhoids in a level III and IV in the Lord scale.

In the surgery Longo's intervention would be done by two ways differing in the distance of the suture from the tobacco pouch to the anal margin (4.5 cm in the first group and 6 cm in the second group).

ELIGIBILITY:
Inclusion Criteria:

* Women and men from 18 to 70 years old
* Hemorrhoids in level III and IV in the Lord scale
* Surgery without income and conventional hospitalization

Exclusion Criteria:

* Previous hemorrhoidal intervention
* Actual anal pathology

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2004-04-04 (Actual); Primary Completion 2012-02-29 (Actual); Study Completion 2012-02-29 (Actual)

PRIMARY OUTCOMES:
Efficacy of the Longo's intervention (distance in the staple line till the dentate line of the anal canal in cm) | up to 6 months
  The distance in the staple line till the dentate line of the anal canal will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Lluis Hidalgo, Principal Investigator — Hospital de Mataró
Locations (1):
- Hospital de Mataró, Mataró, Barcelona, Spain

REFERENCES:
- [Derived] Hidalgo-Grau LA, Piedrafita-Serra E, Ruiz-Edo N, Llorca-Cardenosa S, Heredia-Budo A, Estrada-Ferrer O, Sunol-Sala X. Prospective Randomized Study on Stapled Anopexy Height and Its Influence on Recurrence for Hemorrhoidal Disease Treatment. World J Surg. 2020 Nov;44(11):3936-3942. doi: 10.1007/s00268-020-05676-y. PMID 32647985